CLINICAL TRIAL: NCT02810652
Title: Perioperative Geriatrics Intervention for Older Cancer Patients Undergoing Surgical Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Ryan Nipp, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-189
Record Dates: First submitted 2016-06-16; First posted 2016-06-23 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Pancreatic Cancer; Esophageal Cancer; Gastric Cancer; Rectal Cancer; Hepatobiliary Cancer; Colon Cancer
Keywords: Cancer Surgery Care
MeSH Terms: conditions — Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Rectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perioperative Geriatrics Intervention (Experimental): Evaluation with a board-certified geriatric clinician, both pre- and post-operatively.
  Interventions: Other: Perioperative Geriatrics Intervention
- Standard Care (Active Comparator): Usual care participants will not meet with a geriatric clinician perioperatively, but may receive a geriatric consult upon request or at the discretion of their treating clinician(s).
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Usual Care — Usual Care participants will not meet with a geriatric clinician perioperatively, though they may receive a geriatric consult at their request or at the discretion of their treating cancer team.
  Arms: Standard Care
Other: Perioperative Geriatrics Intervention — Patients randomized to the perioperative geriatrics intervention will undergo evaluation with a board-certified Massachusetts General Hospital (MGH) geriatric clinician, both pre- and post-operatively. The geriatric clinician visits will focus on the following issues: comorbidity, polypharmacy, nutrition, physical and mental function, and social support.
  Arms: Perioperative Geriatrics Intervention

SUMMARY:
The purpose of this research study is to addresses the challenge of managing the unique perioperative needs of older cancer patients undergoing surgical resection.

DETAILED DESCRIPTION:
In the proposed study, the investigators will conduct a randomized controlled trial of a perioperative geriatrics intervention versus usual care in older patients with gastrointestinal (GI) cancers undergoing surgical resection. The perioperative geriatrics intervention will entail pre- and post-operative geriatric care for patients age ≥65 undergoing surgery for gastrointestinal cancers. Specifically, geriatric clinicians will evaluate and manage patients preoperatively in the outpatient setting and postoperatively in the inpatient setting as a consultant.

The investigators will evaluate the effect of the perioperative geriatrics intervention on postoperative length of stay (primary outcome) and readmissions in a sample of 160 patients. The investigators will also assess the impact of the perioperative geriatrics intervention on patient-reported outcomes, including quality of life (QOL) and symptom burden.

The study will take place at Massachusetts General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Diagnosed with pancreatic, esophageal, rectal, colon, hepatobiliary, or gastric cancer (including patients with prior diagnosis of another cancer)
* Planning to receive surgical resection at MGH (including both curative and palliative resections)
* Verbal fluency in English

Exclusion Criteria:

* Unwilling or unable to participate in the study
* Significant uncontrolled psychiatric disorder (e.g. psychotic disorder, bipolar disorder, major depression) or other co-morbid disease (e.g. dementia, cognitive impairment) which the treating clinician believes prohibits informed consent or participation in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-09; Primary Completion 2020-09 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Hospital Length Of Stay | 2 years
  Hospital length of stay from admission to discharge

SECONDARY OUTCOMES:
30-day readmission rate | 2 years
  Defined as the first hospital readmission within 30 days of prior hospital discharge, if patients are readmitted
Time to readmission | 2 years
  Defined as time from discharge to first readmission.
Change In patients' QOL From Baseline To Post-Intervention | For all patient-reported outcomes, change from baseline to post-intervention is defined as change from baseline to post-operative day 5 (±1 day) and from baseline to post-operative day 30 (±7 days)]
  For all patient-reported outcomes, change from baseline to post-intervention is defined as change from baseline to post-operative day 5 (±1 day) and from baseline to post-operative day 30 (±7 days)]
Change In Patients' Symptom Scores From Baseline To Post-Intervention | For all patient-reported outcomes, change from baseline to post-intervention is defined as change from baseline to post-operative day 5 (±1 day) and from baseline to post-operative day 30 (±7 days)]
  Edmonton Symptom Assessment System (ESAS) symptom scores measured continuously
Change In Patients' Depression From Baseline To Post-Intervention | For all patient-reported outcomes, change from baseline to post-intervention is defined as change from baseline to post-operative day 5 (±1 day) and from baseline to post-operative day 30 (±7 days)]
  As per Geriatric Depression Scale (GDS) measured continuously
Rates Of Post-Intervention Depression Symptoms | For all patient-reported outcomes, change from baseline to post-intervention is defined as change from baseline to post-operative day 5 (±1 day) and from baseline to post-operative day 30 (±7 days)]
  Defined as presence of GDS scores > 5
Rates Of Post-Intervention Moderate/Severe Symptoms | For all patient-reported outcomes, change from baseline to post-intervention is defined as change from baseline to post-operative day 5 (±1 day) and from baseline to post-operative day 30 (±7 days)]
  Defined as presence of Edmonton Symptom Assessment System (ESAS) scores ≥4
Change In Activities of Daily Living (ADLs) / Instrumental Activities of Daily Living (IADLs) From Baseline To Post-Intervention | For all patient-reported outcomes, change from baseline to post-intervention is defined as change from baseline to post-operative day 5 (±1 day) and from baseline to post-operative day 30 (±7 days)]
  As per the Medical Outcomes Study (MOS) and the Older American Resources and Services (OARS) measured continuously
Change In The Number Of Falls During The Past 6 Months (measured continuously) From Baseline To Post-Intervention. | For all patient-reported outcomes, change from baseline to post-intervention is defined as change from baseline to post-operative day 5 (±1 day) and from baseline to post-operative day 30 (±7 days)]
  Patient self-report of falls
Rates Of Post-Intervention Activity of Daily Living (ADL) Deficits | For all patient-reported outcomes, change from baseline to post-intervention is defined as change from baseline to post-operative day 5 (±1 day) and from baseline to post-operative day 30 (±7 days)]
  Defined as presence of any Activity of Daily Living (ADL) deficit
Rates Of Post-Intervention Instrumental Activity of Daily Living (IADL) Deficits | For all patient-reported outcomes, change from baseline to post-intervention is defined as change from baseline to post-operative day 5 (±1 day) and from baseline to post-operative day 30 (±7 days)]
  Defined as presence of any Instrumental Activity of Daily Living (IADL) deficit
Rates Of Post-Intervention Falls | For all patient-reported outcomes, change from baseline to post-intervention is defined as change from baseline to post-operative day 5 (±1 day) and from baseline to post-operative day 30 (±7 days)]
  Defined as presence of any falls

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Nipp, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No